CLINICAL TRIAL: NCT03480789
Title: the Influence of Sleep Improvement Through Different Methods on Patients in ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sleep in ICU
Record Dates: First submitted 2018-03-18; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-01

CONDITIONS: Metabolic Problems; Sleep
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- eye patch (Experimental): wearing the eye patch from 22:00 to 6:00 of the next day
  Interventions: Device: eye patch
- Dexmedetomidine (Experimental): given dexmedetomidine to meet RASS -1 from 22:00 to 6:00 of the next day
  Interventions: Drug: Dexmedetomidine
- eye patch + DEX (Experimental): given dexmedetomidine to meet RASS -1 and wearing the eye patch from 22:00 to 6:00 of the next day
  Interventions: Drug: Dexmedetomidine; Device: eye patch
- usual treatment (No Intervention): treatment as usual

INTERVENTIONS:
Drug: Dexmedetomidine — given dexmedetomidine to meet RASS -1 from 22:00 to 6:00 of the next day
  Other Names: Precedex
  Arms: Dexmedetomidine; eye patch + DEX
Device: eye patch — wearing the eye patch from 22:00 to 6:00 of the next day
  Other Names: blinders
  Arms: eye patch; eye patch + DEX

SUMMARY:
In the research, we enroll 120 postoperative patients in the ICU and they will be assigned to four group: the eye patch group, the Dexmedetomidine(DEX) group, the eye patch+DEX group and the usual group. The sleep quality would be evaluated by the EEG monitor and the metabolic level, the inflammation and nutrition status would be detected.

DETAILED DESCRIPTION:
In the research, we enroll 120 postoperative patients in the ICU and they will be assigned to four group: the eye patch group, the Dexmedetomidine(DEX) group, the eye patch+DEX group and the usual group. The sleep quality would be evaluated by the EEG monitor and the metabolic level, the inflammation and nutrition status would be detected. The research aims to confirm that the sleep quality could have a great influence on patients in the ICU and different interventions would make various changes.

ELIGIBILITY:
Inclusion Criteria:

* the postoperative patients that admission to icu is more than 48h

Exclusion Criteria:

* pregnant or breastfeeding
* sleep disorders before operation
* poor liver or kidney function
* post craniocerebral operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-31 (Estimated)

PRIMARY OUTCOMES:
the total time of sleep | the first 24hours in the icu
  using EEG records the time of sleep and different sleep phases

CONTACTS AND LOCATIONS:
Locations (1):
- The Affliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu, China